CLINICAL TRIAL: NCT03914157
Title: Ultrasound Wave Therapy for Post-stenotic Microvascular Remodeling
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to support study
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rajiv Gulati, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-007617; R01HL123160 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Intervention Model Description: We will study 30 patients with ARAS randomized to SWT or sham (n=15 each) twice a week over 3 weeks. We will measure before and again 3 months after a 3-wk regimen renal cortical and medullary perfusion and function (multi-detector computed tomography [MDCT]), oxygenation, and fibrosis (magnetic resonance imaging [MRI]), urinary and plasma levels of renal injury markers, systemic endothelial function, and heart rate variability, an index of sympathetic activation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 15 patients with ARAS randomized to SWT (Active Comparator): We will study 15 patients with ARAS randomized to SWT twice a week over 3 weeks. We will measure before and again 3 months after a 3-wk regimen renal cortical and medullary perfusion and function (multi-detector computed tomography [MDCT]), oxygenation, and fibrosis (magnetic resonance imaging [MRI]), urinary and plasma levels of renal injury markers, systemic endothelial function, and heart rate variability, an index of sympathetic activation.
  Interventions: Device: Low-energy extracorporeal ultrasound shockwave therapy (SWT)
- 15 patients with ARAS sham (Sham Comparator): we will study 15 patients with ARAS randomized to or sham twice a week over 3 weeks. We will measure before and again 3 months after a 3-wk regimen renal cortical and medullary perfusion and function (multi-detector computed tomography [MDCT]), oxygenation, and fibrosis (magnetic resonance imaging [MRI]), urinary and plasma levels of renal injury markers, systemic endothelial function, and heart rate variability, an index of sympathetic activation.
  Interventions: Device: Low-energy extracorporeal ultrasound shockwave therapy (SWT)

INTERVENTIONS:
Device: Low-energy extracorporeal ultrasound shockwave therapy (SWT) — SWT delivers 10% energy of the traditional SWT used for clinically indicated lithotripsy, evokes neovascularization, and improves regional blood flow and function in various ischemic tissues.

SUMMARY:
Researchers are evaluating a noninvasive treatment with ultrasound waves for Atherosclerotic Renal Artery Stenosis (ARAS).

DETAILED DESCRIPTION:
Investigators will study 30 patients with ARAS randomized to SWT or sham (n=15 each) twice a week over 3 weeks. We will measure before and again 3 months after a 3-wk regimen renal cortical and medullary perfusion and function (multi-detector computed tomography [MDCT]), oxygenation, and fibrosis (magnetic resonance imaging [MRI]), urinary and plasma levels of renal injury markers, systemic endothelial function, and heart rate variability, an index of sympathetic activation.

ELIGIBILITY:
Inclusion Criteria

* Patients are between ages 40 and 80 years old.
* Patients with hypertension (Systolic BP> 155 mm Hg) and/or requirement for two or more antihypertensive medications for more than 4 weeks, no restrictions on antihypertensive agents, although loop diuretics may be changed to diluting site agents (e.g. hydrochlorothiazide, indapamide, metolazone) for two weeks prior to study.
* Patients have serum creatinine ≤2.2 mg/dL.
* Patients have no contraindications to angiography: severe contrast allergy.
* Patients have no contraindications to no-contrast MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia.
* Patients have the ability to comply with protocol
* Patients are competent and able to provide written informed consent

Exclusion Criteria

* Patient have serum creatinine >2.2 mg/dL
* ARAS in a solitary kidney
* Patients have clinically significant medical conditions within the six months before SWT treatment: e.g. myocardial infarction, congestive heart failure, stroke, that would, in the opinion of the investigators, compromise the safety of the patient.
* Uncontrolled hypertension (Systolic BP >180 mmHg despite therapy).
* Pacemaker, implantable defibrillator or other contraindication to MRI
* Inability to comply with breath-hold for 20 seconds
* Any active malignancy and undergoing therapy
* Patients are pregnant.
* Kidney or ureteric stone that may affect the effect of SWT.
* Another known acute or chronic kidney disease
* Local inflammation or infection over treatment areas.
* Bleeding disorders.
* Federal medical center inmates.
* Latex allergy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in kidney perfusion assessed by computed tomography | Baseline, 3 months
  Single-kidney perfusion and GFR assessed by multi-detector computed tomography (MDCT)
Change in renal function assessed by GFR | Baseline, 3 months
  Renal function by eGFR calculated by both the modified modification of Diet in Renal Disease (MDRD) formula, and measured GFR (mGFR) by iothalamate clearance
Change in blood oxygen in kidney assessed by MRI | Baseline, 3 months
  Cortical and medullary oxygenation assessed by Blood oxygen-level-dependent (BOLD)-MRI
Change in renal fibrosis assessed by MRI | Baseline, 3 months
  Renal fibrosis as determined by Magnetization transfer imaging (MTI)-MRI in vivo.
Change in urinary levels of biomarkers and extracellular vehicles | Baseline, 3 months
  Urinary biomarkers albumin, renal injury markers: Neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecular (KIM)-1, and lactate dehydrogenase (LDH)], as well as urinary levels of extracellular vehicles (EVs) (measured by flow cytometry) originating from renal microvessels.
Change in labs collected from right and left renal veins and/or Inferior Vena Cava | Baseline, 3 months
  Serum creatinine, plasma renin activity (PRA), aldosterone, cytokines and circulating endothelial progenitor cell (EPC) in blood collected from the left and right renal veins and the Inferior Vena Cava (IVC).
Change in mean arterial pressure assessed by oscillometry | Baseline, 3 months
  systolic and diastolic BP will be measured by oscillometry to calculate MAP, and assessment of sympathetic nervous system activation by heart rate variability (HRV).
Change in peripheral microvascular endothelial function assessed in the fingertip | Baseline, 3 months
  Peripheral microvascular endothelial function by peripheral arterial tonometry (EndoPAT).

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Gulati, MD, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No
We do not intend to make individual participant data (IPD) available to other researchers.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials